CLINICAL TRIAL: NCT05505682
Title: Assessing the Efficacy of Male Wolbachia-infected Mosquito Deployments to Reduce Dengue Incidence in Singapore: a Cluster Randomized Controlled Trial
Brief Title: Impact of Project Wolbachia - Singapore on Dengue Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Environment Agency, Singapore (Other Government)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Lee Ching Ng, Group Director (Environmental Health Institute), National Environment Agency, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB024
Record Dates: First submitted 2022-07-19; First posted 2022-08-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: Parallel, two-arm, non-blinded cluster-randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention clusters (Experimental): Residential areas that receive releases of male Wolbachia-infected Aedes aegypti
  Interventions: Biological: Biological (Male Wolbachia-infected Aedes aegypti)
- Non-intervention clusters (No Intervention): Residential areas that do not receive releases of male Wolbachia-infected Aedes aegypti

INTERVENTIONS:
Biological: Biological (Male Wolbachia-infected Aedes aegypti) — Releases of male Wolbachia-infected Aedes aegypti mosquitoes
  Arms: Intervention clusters

SUMMARY:
The study is a cluster-randomised controlled trial set in Singapore, to assess if the deployment of male Wolbachia-infected Aedes aegypti mosquitoes can reduce dengue incidence in intervention clusters.

DETAILED DESCRIPTION:
The study is designed as a parallel, two-arm, non-blinded cluster-randomised controlled trial to be conducted in high-rise public housing estates in Singapore. The aim is to determine whether large-scale deployment of male Wolbachia-infected Ae. aegypti mosquitoes can significantly reduce dengue incidence in intervention clusters. The investigators will use the cluster-randomised design, with the study area comprising 15 clusters with a total area of 10.9 km2, covering approximately 722,000 residents in 1,700 apartment blocks. Eight clusters will be randomly selected to receive the intervention, while the other seven will serve as non-intervention clusters. Intervention efficacy will be estimated through two primary endpoints: (1) odds ratio of Wolbachia exposure distribution (i.e. probability of living in an intervention cluster) among laboratory-confirmed reported dengue cases compared to test-negative controls, and (2) laboratory-confirmed reported dengue counts normalized by population size in intervention versus non-intervention clusters.

ELIGIBILITY:
Inclusion criteria:

* Dengue-suspected patients living in the intervention and non-intervention clusters whose blood samples are collected by a national network of diagnostic laboratories that support private clinics, public polyclinics, or public/private hospitals.
* Test positive cases: Patients with virologically confirmed DENV infection through RT-qPCR, testing positive for NS1 antigen or IgM. A positive test for any of the three assays would classify the patient as a dengue case.
* Test negative controls: Patients with negative test results for DENV through RT-qPCR, NS1 antigen ELISA, or DENV IgM.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 724428 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Odds ratio of Wolbachia exposure distribution among laboratory-confirmed reported dengue cases compared to test-negative controls | Up to 3 years
  Dengue cases and dengue test-negative controls data will be obtained from the national surveillance network of diagnostic laboratories which receive samples for dengue testing.
Laboratory-confirmed reported dengue case counts normalized by population size in intervention versus non-intervention clusters | Up to 3 years
  Dengue cases data will be obtained from the national surveillance network of diagnostic laboratories which receive samples for dengue testing.

SECONDARY OUTCOMES:
Prevalence of Ae. aegypti/Ae. albopictus mosquitoes | Up to 3 years
  Data will be obtained from the national gravitrap surveillance system
Public Attitudes, Perceptions & Knowledge (APK) of Wolbachia and other vector control interventions | Up to 3 years
  Sentiment surveys pre-trial and during the course of the trial, using true/false and Likert-type scales. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ching Ng, PhD, Principal Investigator — Group Director (Environmental Health Institute)
Locations (1):
- National Environment Agency, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anders KL, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Andari B, Jewell NP, Rances E, O'Neill SL, Simmons CP, Utarini A. The AWED trial (Applying Wolbachia to Eliminate Dengue) to assess the efficacy of Wolbachia-infected mosquito deployments to reduce dengue incidence in Yogyakarta, Indonesia: study protocol for a cluster randomised controlled trial. Trials. 2018 May 31;19(1):302. doi: 10.1186/s13063-018-2670-z. PMID 29855331
- [Background] Utarini A, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Ansari MR, Supriyati E, Wardana DS, Meitika Y, Ernesia I, Nurhayati I, Prabowo E, Andari B, Green BR, Hodgson L, Cutcher Z, Rances E, Ryan PA, O'Neill SL, Dufault SM, Tanamas SK, Jewell NP, Anders KL, Simmons CP; AWED Study Group. Efficacy of Wolbachia-Infected Mosquito Deployments for the Control of Dengue. N Engl J Med. 2021 Jun 10;384(23):2177-2186. doi: 10.1056/NEJMoa2030243. PMID 34107180
- [Derived] Lim JT, Mailepessov D, Chong CS, Chang CC, Dickens B, Lai YL, Deng L, Lee C, Tan LY, Chain G, Ho SH, Zulkifli MF, Liew J, Vasquez K, Lee V, Wong JCC, Sim S, Tan CH, Ng LC. Update to: Assessing the efficacy of male Wolbachia-infected mosquito deployments to reduce dengue incidence in Singapore. Trials. 2024 Jun 20;25(1):400. doi: 10.1186/s13063-024-08148-z. PMID 38902790
- [Derived] Ong J, Ho SH, Soh SXH, Wong Y, Ng Y, Vasquez K, Lai YL, Setoh YX, Chong CS, Lee V, Wong JCC, Tan CH, Sim S, Ng LC, Lim JT. Assessing the efficacy of male Wolbachia-infected mosquito deployments to reduce dengue incidence in Singapore: study protocol for a cluster-randomized controlled trial. Trials. 2022 Dec 17;23(1):1023. doi: 10.1186/s13063-022-06976-5. PMID 36528590